CLINICAL TRIAL: NCT00380523
Title: Analgesic Treatment Mediated by Arcoxia
Brief Title: Analgesic Treatment Mediated by Arcoxia (0663-093)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0663-093; 2006_034
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Etoricoxib; Duration of Therapy

INTERVENTIONS:
Drug: MK0663, Arcoxia, etoricoxib / Duration of Treatment: 3 Days

SUMMARY:
Allow physicians to test the efficacy of arcoxia in patients with acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pain susceptible of pharmacological treatment
* Greater than 18 years of age
* Voluntary acceptance to participate in the study and signature of the informed consent form

Exclusion Criteria:

* Allergy to etoricoxib or any of its components
* Less than 18 years old
* Patient is taking anticoagulants
* Patient that already has taken any drug as analgesic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2005-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Evaluate pain using the verbal analog scale (evaluate pain before starting treatment and then evaluate pain every day after had taken arcoxia up to three days)

SECONDARY OUTCOMES:
Patient satisfaction with the drug therapy using PGART scale
Patient satisfaction was obtained at the end of treatment(on third day)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC